CLINICAL TRIAL: NCT00001614
Title: The Safety and Efficacy of Chicken Type II Collagen on Uveitis Associated With Juvenile Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970146; 97-EI-0146
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Arthritis, Juvenile Rheumatoid; Uveitis
Keywords: Eye; Immunosuppression; Inflammation; Iritis; Joint; Oral Tolerance; Juvenile Rheumatoid Arthritis; Uveitis
MeSH Terms: conditions — Arthritis, Juvenile; Uveitis; Inflammation; Iritis

INTERVENTIONS:
Drug: Chicken type II collagen

SUMMARY:
Current treatment modalities for uveitis associated with juvenile rheumatoid arthritis have not been beneficial in the juvenile population. A new approach for treating patients with presumed autoimmune disorders is oral tolerance therapy. Chicken type II collagen (Colloral) is being developed as an oral tolerance therapy for the treatment of rheumatoid arthritis. This open label pilot study will describe the safety of chicken type II collagen added to current anti-inflammatory medications as treatment for patients with uveitis associated with juvenile rheumatoid arthritis. The primary ophthalmic outcomes of this study will be a change from baseline in the number of anterior chamber cells and the number and dosage of anti-inflammatory medications. Secondary outcomes for JRA will include change in physician's global assessment, parent/patient assessment of overall well-being, functional assessment, number of joints with active arthritis, number of joints with limited range of motion, and erythrocyte sedimentation rate (ESR). Secondary outcomes for uveitis will include change in visual acuity, vitreous haze, and anterior chamber flare.

DETAILED DESCRIPTION:
Current treatment modalities for uveitis associated with juvenile rheumatoid arthritis have not been beneficial in the juvenile population. A new approach for treating patients with presumed autoimmune disorders is oral tolerance therapy. Chicken type II collagen (Colloral) is being developed as an oral tolerance therapy for the treatment of rheumatoid arthritis. This open label pilot study will describe the safety of chicken type II collagen added to current anti-inflammatory medications as treatment for patients with uveitis associated with juvenile rheumatoid arthritis. The primary ophthalmic outcomes of this study will be a change from baseline in the number of anterior chamber cells and the number and dosage of anti-inflammatory medications. Secondary outcomes for JRA will include change in physician's global assessment, parent/patient assessment of overall well-being, functional assessment, number of joints with active arthritis, number of joints with limited range of motion, and erythrocyte sedimentation rate (ESR). Secondary outcomes for uveitis will include change in visual acuity, vitreous haze, and anterior chamber flare.

ELIGIBILITY:
Must meet American College of Rheumatology Criteria for JRA.

Must have active anterior uveitis defined as the presence of inflammatory cells in the anterior chamber in at least one eye, or the current use of topical corticosteroids.

Must be between 2 and 18 years of age, inclusive.

Must have had previous therapy for uveitis.

Must be able to undergo a slit lamp biomicroscopy for assessment of anterior chamber cells.

Must not have a media opacity that precludes assessment of anterior chamber inflammation.

Must not have received a periocular injection of corticosteroids within 2 months of baseline.

Must not be currently receiving DMARD (disease modifying anti-rheumatic) therapy, with the exception of prednisone at a dose no greater than 1.5-2.0 mg/kg/day, or methotrexate at a dose no greater than 10 mg/m(2)/week.

Must not have active eye or joint inflammation requiring immediate addition or increase in systemic anti-inflammatory medications.

Must not have involvement in prior clinical trials of type II collagen.

Must not have exposure within the past year to shark or other collagen preparations found in health food stores.

Must not have a history of gastrointestinal disease which could affect the presentation of type II collagen.

Women must not be pregnant or lactating.

Patients currently using Latanoprost, patients who have used Latanoprost within the last 2 weeks, or patients who are likely to need Latanoprost during the course of the study will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13
Dates: Start 1997-07; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Trentham DE, Dynesius-Trentham RA, Orav EJ, Combitchi D, Lorenzo C, Sewell KL, Hafler DA, Weiner HL. Effects of oral administration of type II collagen on rheumatoid arthritis. Science. 1993 Sep 24;261(5129):1727-30. doi: 10.1126/science.8378772.
- [Background] Rosenberg AM. Uveitis associated with juvenile rheumatoid arthritis. Semin Arthritis Rheum. 1987 Feb;16(3):158-73. doi: 10.1016/0049-0172(87)90019-9. PMID 3547655